CLINICAL TRIAL: NCT00811525
Title: Post Approval Continued Access Study of the MENTOR® Contour Profile Gel Breast Implant
Acronym: CPG-CA
Status: Approved for marketing | Type: Expanded Access
Sponsor: Mentor Worldwide, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 110390CA-0912-2
Record Dates: First submitted 2008-12-17; First posted 2008-12-19 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Breast Augmentation; Breast Reconstruction; Breast Revision
Keywords: Breast Augmentation; Breast Reconstruction; Breast Revision; Silicone gel; Contour Profile Gel; Siltex

INTERVENTIONS:
Device: Mentor Siltex® Contour Profile Gel Mammary Prosthesis — The CPG mammary prosthesis is a silicone elastomer mammary device with a textured surface. The Siltex® (textured) shell consists of a smooth shell bonded to an additional layer of silicone that has a textured pattern imprinted into its surface. The Siltex® shell is textured to provide a disruptive surface for collagen interface. The CPG implant contains a gel that is a more cohesive silicone gel than that used in other Mentor gel implants. The gel is made from the same materials as Mentor's standard gel. The contour shape of the CPG is designed to provide inferior projection with reduced superior fullness. The CPG mammary prosthesis contains raised orientation marks on the anterior and posterior of the implant which may help the physician ensure proper placement. CPG was available in sizes 120 cc-775 cc and 5 styles with various projection and height options.
  With approval of MemoryShape™ (CPG 321) Breast Implants, the study converted to a post approval study for this style.
  Other Names: MemoryShape™ Breast Implants

SUMMARY:
The Contour Profile Gel Continued Access Study is designed to demonstrate safety of Mentor's Mammary Prostheses in women who are undergoing primary augmentation, primary reconstruction, or revision. Safety information on the rate of capsular contracture, rupture, and infection will be collected, and used to help determine device safety.

With approval of MemoryShape™ Medium Height, Moderate Profile (CPG 321) Breast Implants on June 14, 2013, CPG CA Study subject enrollment has closed and the study has converted to a post approval study for this style.

DETAILED DESCRIPTION:
Silicone gel-filled breast implants were introduced in the early sixties and were in wide-scale distribution by the time the Medical Device Amendments to the Food Drug and Cosmetic Act was passed in 1976. In 1983, gel-filled breast implants were designated as Class III devices requiring premarket approval. In May 1990, the Food and Drug Administration (FDA) published a proposed request (515(b)) for Premarket Approval Applications (PMA) and in April 1991 published the final request. This final publication put manufacturers of gel-filled breast implants on notice that for continued marketing of gel-filled breast implants, a PMA was due to FDA in 90 days from the final publication date.

A premarket approval (PMA) for the Mentor gel-filled breast implants was filed with the FDA in July 1991. At the FDA General and Plastic Surgery Advisory Committee meeting in November 1991, the committee recommended the submission of additional information to establish the safety and effectiveness of gel-filled breast implants.

In January 1992, the FDA Commissioner announced a voluntary moratorium of the sale of gel-filled breast implants to allow the advisory panel time to assess additional information. In April 1992, the moratorium was lifted but only for reconstruction and revision patients. Every patient implanted had to be part of an adjunct study, and had to be offered participation in a registry of gel-filled breast implant patients. In order to be implanted with gel-filled implants for augmentation, women had to be enrolled in a core clinical study.

In September of 2000 the Core Gel study began, leading the way to the November 2006 FDA approval of the Core Gel implant or Memory Gel breast implant.

The objective of the Contour Profile Gel Continued Access is to determine the safety of the Silicone Contour Profile Gel Mammary Prostheses in women who are undergoing primary breast augmentation, primary breast reconstruction, or revision. While Core CPG patient follow-up is being completed, this Continued Access Study was designed to enroll patients at a limited rate per month to allow for continued physician experience with the device and to collect additional safety data to support a future PMA. Safety data will be collected and submitted as supplemental data. The CPG-CA study includes the same original investigators and surgical sites in the Core CPG study. However, not all of the original Core CPG investigators are in the CPG-CA study.

Throughout the duration of this study, patients are required to have follow-up visits at 10 weeks post-surgery and every year after surgery through the 10th year of completion as in the Core CPG study. (This follow-up requirement changed from 10 years to 5 years upon device approval). Unlike the Core CPG study, the CPG-CA study does not have a randomized selection of MRI patients as a required component of the study.

On June 14, 2013, the FDA approved Mentor® MemoryShape™ Breast Implants (CPG Style 321 Medium Height, Moderate Profile) for the following indications:

* Breast Augmentation for women at least 22 years old.
* Breast Reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Subject is Genetic female and is at least 18 years old
* A candidate for:

  * Primary breast augmentation (for general breast enlargement)
  * Primary breast reconstruction (for cancer, trauma, surgical loss of breast or congenital deformity)
  * Revision surgery (previous augmentation or reconstruction with silicone-filled or saline-filled implants)
* Signs the Informed Consent
* Agrees to return device to Mentor if device is explanted
* Agrees to comply with follow-up procedures, including returning for all follow-up visits

Exclusion Criteria:

* Subject is pregnant
* Has nursed a child within three months of study enrollment
* Been implanted with any silicone implant other than breast implants
* Confirmed diagnosis of rheumatic disease
* Currently has a condition that could compromise or complicate wound healing (except reconstruction subjects)
* Subject in Augmentation cohort and has diagnosis of active cancer of any type, except low-grade non-metastasizing skin cancer
* Infection or abscess anywhere in the body
* Demonstrates tissue characteristics which are clinically incompatible with implant (e.g. tissue damage resulting from radiation, inadequate tissue, or compromised vascularity)
* Possesses any condition, or is under treatment for any condition which, in the opinion of the investigator and/or consulting physicians(s), may constitute an unwarranted surgical risk.
* Anatomic or physiologic abnormality which could lead to significant postoperative adverse events
* Demonstrates characteristics that are unrealistic/unreasonable with the risks involved with the surgical procedure
* Premalignant breast disease without a subcutaneous mastectomy.
* Untreated or inappropriately treated breast malignancy, without mastectomy
* Are HIV positive
* Work for Mentor or the study doctor or are directly-related to anyone that works for Mentor or the study doctor

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Dates: Start 2004-08

CONTACTS AND LOCATIONS:
Overall Officials: William Adams, M.D., Principal Investigator — Dallas, TX; Frank Barone, M.D., Principal Investigator — Toledo, OH; Joseph Bauer, M.D., Principal Investigator — Alpharetta, GA; Michael Bentley, M.D., Principal Investigator — Montgomery, AL; John Bishop, M.D., Principal Investigator — Greenville, SC; David Caplin, M.D., Principal Investigator — St. Louis, MO; E. Dale Collins Vidal, M.D., Principal Investigator — Lebanon, NH (Dartmouth-Hitchcock); Craig Colville, M.D., Principal Investigator — Toledo, OH; Gloria Duda, M.D., Principal Investigator — McLean, VA (D.C. Metro area); Barry Fernando, M.D., Principal Investigator — Phoenix, AZ; William Gorman, M.D., Principal Investigator — Austin, TX; Scot Glasberg, M.D., Principal Investigator — New York, NY; Strawford Dees, M.D., Principal Investigator — Biloxi, MS; Dennis Hammond, M.D., Principal Investigator — Grand Rapids, MI; Mark Jewell, M.D., Principal Investigator — Eugene, OR; Robert Kevitch, M.D., Principal Investigator — Allentown, PA; Shujaat Khan, M.D., Principal Investigator — Fort Worth, TX; Philip Kierney, M.D., Principal Investigator — Puyallup, WA; John Lettieri, M.D., Principal Investigator — Spartanburg, SC; Tim Love, M.D., Principal Investigator — Oklahoma City, OK; Mark Migliori, M.D., Principal Investigator — Edina, MN; Bradley Remington, M.D., Principal Investigator — Kirkland, WA; John Smoot, M.D., Principal Investigator — La Jolla, CA; Grant Stevens, M.D., Principal Investigator — Marina Del Rey, CA; Steven Teitelbaum, M.D., Principal Investigator — Santa Monica, CA; Lewis Berger, M.D., Principal Investigator — Tampa, FL; Patrick Maxwell, M.D., Principal Investigator — Nashville, TN; Jack Fisher, M.D., Principal Investigator — Nashville, TN; David A. Stoker, M.D., Principal Investigator — Marina Del Rey, CA